CLINICAL TRIAL: NCT04901078
Title: A Phase 1 Study Investigating the Safety, Tolerability and Pharmacokinetics of KNX100 in Healthy Volunteers
Acronym: KTX101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kinoxis Therapeutics Pty Ltd (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: KTX101; 1UG3DA048743-01 (NIH)
Record Dates: First submitted 2021-05-09; First posted 2021-05-25 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteer Study; Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Dosing will be based on the assigned treatment group. The single ascending dose cohorts will evaluate doses of KNX100 starting with 25 mg and increasing up to a maximum of 50 mg per day. The multiple ascending dose cohorts will evaluate a low-, mid-, and high-dose KNX100 administered for 7 consecutive days. Individual doses will be dispensed by unblinded site pharmacy staff. Dose escalation will progress upon Cohort Review Committee (CRC) approval.
Who Masked: Participant, Investigator
Masking Description: This will be a double blinded, randomised, placebo study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): KNX100 which will be provided in capsule form as 5, 25 and 100 mg capsules for oral administration. Study drug will be encapsulated in hydroxypropyl methylcellulose (HPMC) dark green opaque size 0 capsules and packaged in 100 mL high density polyethylene (HDPE) bottles with polypropylene (PP) twist-off closures.
  Interventions: Drug: KNX100
- Placebo (Placebo Comparator): KNX100 matching placebo will be provided in capsule form for oral administration. The placebo will be encapsulated in HPMC dark green opaque size 0 capsules and packaged in 100 mL HDPE bottles with PP twist-off closures.
  Interventions: Drug: KNX100

INTERVENTIONS:
Drug: KNX100 — KNX100 will be provided in capsule form as 5, 25 and 100 mg capsules for oral administration. Study drug will be encapsulated in hydroxypropyl methylcellulose (HPMC) dark green opaque size 0 capsules and packaged in 100 mL high density polyethylene (HDPE) bottles with polypropylene (PP) twist-off closures.
  Other Names: KNX100 placebo

SUMMARY:
The primary objectives of this study are to evaluate the safety and tolerability of KNX100 administered orally as a single and multiple ascending doses in healthy volunteers.

DETAILED DESCRIPTION:
This is an adaptive, Phase 1, first-in-human (FIH), single treatment, double blind, placebo controlled, randomized, single and multiple ascending dose study of KNX100 administered to healthy volunteers. Approximately 64 male and female healthy subjects will be enrolled into this study. Healthy subjects who meet all the eligibility criteria will be randomly assigned to Cohorts 1-5 for the Single Ascending Dose and Cohorts 1-3 for the Multiple Ascending Dose. Each cohort will evaluate 8 subjects; 6 subjects will receive KNX100 (study drug) and 2 subjects will receive placebo.

Each cohort will be enrolled sequentially, and dose escalation decisions will be made according to protocol by the Cohort Review Committee (CRC) consisting of the investigators and medical monitor. Subjects and clinical staff will be blinded to therapy assignment. KNX100 will be provided in capsule form as 5, 25 and 100 mg capsules for oral administration and the dose range will be 5 to 50mg.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and provide written informed consent.
2. Body mass index (BMI) within the range of 18-32 (inclusive).
3. Healthy male and female volunteers ≥18 and ≤55 years old at Screening.
4. Able and willing to comply with the requirements of the study and complete the full sequence of protocol related doses, procedures, and evaluations.
5. Willing to agree not to use alcohol or recreational drugs and willing to have drug screening, prior to the first dose of KNX100 and if drug use is suspected while active in the study.
6. Willing to agree not to smoke cigarettes or use tobacco based products prior to the first dose of KNX100 and for the entire duration of the study.
7. Males who are sexually active must use a condom OR be abstinent OR have the same sex partner OR be surgically sterile OR have partner who is of non-childbearing potential, for at least 90 days after the last dose of investigational drug. If female partner is a Woman of Child-Bearing Potential (WOCBP), the female partner must use highly effective methods of contraception, defined as below:

   * Hormonal methods of contraception including oral contraceptives containing combined estrogen and progesterone, a vaginal ring, injectable and implantable hormonal contraceptives, intrauterine hormone-releasing system (e.g., Mirena) and progestogen-only hormonal contraception associated with inhibition of ovulation.
   * Nonhormonal intrauterine device,
   * Bilateral tubal occlusion.

Exclusion Criteria:

1. Clinically significant history or presence of significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, neurological, or psychiatric disorder. Any surgical or medical history which may significantly alter the absorption, metabolism, or elimination of drugs or constitute a risk when taking the study intervention; or interfering with the interpretation of data (e.g., gastric bypass, cyclical vomiting, etc.). This includes a history of lymphoma, leukemia, or any malignancy within 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
2. Subjects who have a sitting or semi-supine blood pressure at screening or Day-1, after resting for at least 3 minutes of systolic blood pressure >140 or <100 mmHg, or diastolic blood pressure >90 or <60 mmHg.
3. Subjects who have a sitting or semi-supine pulse rate at screening or Day-1, after resting for at least 3 minutes, outside the range of <50 or >90 beats/minute
4. Subjects who donated blood or who had a comparable blood loss (approximately 500 mL) during the last 30 days prior to start of this study and while on study.
5. Clinically significant findings on the screening, Day -1, or predose Day 1 electrocardiogram (ECG) or physical examination, including QTcF duration >450 ms for males and >470 ms for females on ECG.
6. Thyroid function tests outside the normal reference ranges and deemed clinically significant by the study PI (and upon repeat).
7. Safety laboratory tests that are outside the normal reference ranges and deemed clinically significant by the study PI (and upon repeat).
8. Any history of meningitis, septicemia, or pneumonia.
9. Any history or family history (first or second degree relative) of seizure disorder, febrile convulsions.
10. Any clinically significant medical history of closed head trauma.
11. Any history of anaphylaxis or other significant allergy.
12. Any current diagnosis or clinically significant medical history of psychiatric illness as diagnosed and documented by a medical practitioner and as defined by the American Psychiatric Association Diagnostic and statistical manual of mental disorders 5th edition (DSM-5).
13. Subjects with a history of chronic alcohol (regular daily intake of more than three standard drinks) or drug abuse within the last 6 months prior to first administration, or evidence of such abuse as indicated by the laboratory profile conducted during the screening examination.
14. Subjects who have received prescription drugs or over-the-counter (OTC) medication including dietary supplements, COVID-19 vaccine, standard dose vitamins, or herbal products within 14 days prior to the first administration (with the exception of the oral contraceptive pill).
15. Subjects who received any treatment agents known to alter the major organs or systems within 30 days prior to the first administration (e.g., diuretics, nephro- or liver toxic medication, barbiturates, phenothiazines, cimetidine, more than 1.0 L of caffeine-containing beverages per day, etc.).
16. Diagnosed infection of any kind, e.g., viral, bacterial, fungal, or mycobacterial within 1 month prior to the first dose of KNX100 or current fever or clinical signs or symptoms of infection at screening or Day -1.
17. Treatment with an unapproved investigational therapeutic agent within 30 days (or 5 half-lives for small molecule agents) prior to the first dose of KNX100.
18. Females who are pregnant (positive pregnancy test at screening or prior to first dose), lactating or unable/unwilling to use defined methods of contraception throughout the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina Soulis, PhD, Study Director — Kinoxis Therapeutics Pty Ltd
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SAD Cohort 1: Part A (SAD) cohort 1 was administered a single dose of 5mg KNX100 capsule.
- SAD- Placebo Cohort: A matching number of placebo capsules were administered per cohort.
- SAD Cohort 2: Part A (SAD) cohort 2 was administered a single dose of 3 x 5mg KNX100 capsules (15mg).
- SAD Cohort 3: Part A (SAD) cohort 3 was administered a single dose of 25mg KNX100 capsule.
- SAD Cohort 4: Part A (SAD) cohort 4 was administered a single dose of 2 X 25mg KNX100 capsules (50mg).
- MAD Cohort 1: Part B(MAD) cohort 1 was administered of 2 x 5mg KNX100 capsules (10mg) once daily for 7 days.
- MAD Cohort 2: Part B (MAD) cohort 2 was administered of 1 x 5mg and 1 x 25mg KNX100 capsules (30mg) once daily for 7 days.
- MAD Cohort 3: Part B (MAD) cohort 3 was administered of 1 x 5mg and 1 x 25mg KNX100 capsules (30mg) twice daily for 7 days.
- MAD-Placebo Cohort: A matching number of placebo capsules were administered for 7 days per cohort.
Period: Overall Study
Arm/Group | SAD Cohort 1 | SAD- Placebo Cohort | SAD Cohort 2 | SAD Cohort 3 | SAD Cohort 4 | MAD Cohort 1 | MAD Cohort 2 | MAD Cohort 3 | MAD-Placebo Cohort
Started | 6 | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SAD Placebo Cohort: Part A (SAD) A single dose of a matching number of placebo capsules were administered per cohort.
- SAD Cohort 2: Part A (SAD) cohort 2 was administered a single dose of 15mg (3 x 5mg) KNX100 capsules.
- SAD Cohort 4: Part A (SAD) cohort 3 was administered a single dose of 50mg (2 x 25mg) KNX100 capsules.
- MAD Placebo Cohort: Part B (MAD) A matching number of placebo capsules were administered either once or twice daily for 7 days.
- MAD Cohort 1: Part B (MAD) cohort 1 was administered of 2 x 5mg KNX100 capsules (10mg) once daily for 7 days.
- MAD Cohort 2: Part B (MAD) cohort 1 was administered of 1 x 5mg and 1x 25mg KNX100 capsules (30mg) once daily for 7 days.
- MAD Cohort 3: Part B (MAD) cohort 1 was administered of 1 x 5mg and 1x 25mg KNX100 capsules (30mg) twice daily for 7 days.
- Total: Total of all reporting groups
Arm/Group | SAD Cohort 1 | SAD Placebo Cohort | SAD Cohort 2 | SAD Cohort 3 | SAD Cohort 4 | MAD Placebo Cohort | MAD Cohort 1 | MAD Cohort 2 | MAD Cohort 3 | Total
Number analyzed (Participants) | 6 | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 56
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (6.06) | 27.6 (8.02) | 29.8 (8.30) | 27.5 (7.01) | 28.2 (8.08) | 32.2 (10.50) | 31.7 (3.72) | 28.3 (3.72) | 27.7 (5.68) | 29.7 (6.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 3 | 2 | 2 | 4 | 2 | 2 | 0 | 24
  Male | 1 | 4 | 3 | 4 | 4 | 2 | 4 | 4 | 6 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 7
  Not Hispanic or Latino | 5 | 7 | 6 | 4 | 6 | 5 | 6 | 6 | 4 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
  Asian | 1 | 3 | 2 | 3 | 2 | 2 | 2 | 0 | 0 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 4 | 4 | 3 | 4 | 3 | 4 | 6 | 5 | 37
  More than one race | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 6 | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 56

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With TEAEs
Description: • Incidence of reported Treatment Emergent Adverse Events (TEAEs), related AEs, AEs leading to discontinuation, and AEs by severity.
Time Frame: From first dose of study drug up to 9 days for SAD cohorts and up to 16 days for MAD cohorts.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo -SAD Cohort: A single dose of matching placebo capsules were administered per cohort.
- SAD Cohort 3: Part A (SAD) cohort 3 was administered a single dose of 25 mg KNX100 capsule.
- SAD Cohort 4: Part A (SAD) cohort 4 was administered a single dose of 50mg (2 x 25mg) KNX100 capsules.
- Placebo - MAD Cohort: Matching placebo capsules were administered once or twice daily per cohort.
Arm/Group | SAD Cohort 1 | Placebo -SAD Cohort | SAD Cohort 2 | SAD Cohort 3 | SAD Cohort 4 | MAD Cohort 1 | MAD Cohort 2 | MAD Cohort 3 | Placebo - MAD Cohort
Number analyzed (Participants) | 6 | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 1 | 1 | 2 | 0 | 3 | 6 | 3 | 4 | 3

ADVERSE EVENTS:
Time Frame: Data collection for Adverse events were collected from the first dose for 24h hours to last dose in clinic, and up to 9 days for SAD cohorts, and up to 16 days for MAD cohorts.
Description: Adverse events were grouped by system organ class (SOC) and preferred term (PT) and summarized by treatment. Treatment-emergent AEs were defined as any AE that started or worsened after the first dose of the study drug.
Groups:
- Placebo SAD Cohort: A single dose of matching placebo capsules were administered per cohort.
- SAD Cohort 2: Part A (SAD) cohort 2 was administered a single dose of 15mg (3 x 5mg) KNX100 capsule.
- SAD Cohort 4: Part A (SAD) cohort 4 was administered a single dose of 50mg (2 x 25mg) KNX100 capsule.
- MAD Cohort 2: Part B (MAD) cohort 2 was administered of 30mg (1 X 25mg + 1 x 5mg) KNX100 capsules once daily for 7 days.
- MAD Cohort 3: Part B (MAD) cohort 2 was administered of 30mg (1 X 25mg + 1 x 5mg) KNX100 capsules twice daily for 7 days.
- Placebo MAD Cohort: Matching placebo capsules were administered once or twice daily per cohort.
Arm/Group | SAD Cohort 1 | Placebo SAD Cohort | SAD Cohort 2 | SAD Cohort 3 | SAD Cohort 4 | MAD Cohort 1 | MAD Cohort 2 | MAD Cohort 3 | Placebo MAD Cohort
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 1/8 | 2/6 | 0/6 | 3/6 | 6/6 | 3/6 | 4/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAD Cohort 1 (N=6) | Placebo SAD Cohort (N=8) | SAD Cohort 2 (N=6) | SAD Cohort 3 (N=6) | SAD Cohort 4 (N=6) | MAD Cohort 1 (N=6) | MAD Cohort 2 (N=6) | MAD Cohort 3 (N=6) | Placebo MAD Cohort (N=6)
somnolence (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Fatique (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site dermatitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Application site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT04901078/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT04901078/SAP_001.pdf